CLINICAL TRIAL: NCT04083911
Title: A Phase 3, Open Label, Single Arm, Multi-Center Study to Evaluate the Efficacy and Safety of Decitabine Combined With HAAG Regimen in Elderly Newly Diagnosed Acute Myeloid Leukemia Patients.
Brief Title: Study of DAC Combined With HAAG Regimen in Newly Diagnosed AML Patients Older Than 60
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: Second Affiliated Hospital of Soochow University (Other); Changzhou No.2 People's Hospital (Other); The First People's Hospital of Lianyungang (Other); Jingjiang People's Hospital (Other); Zhangjiagang First People's Hospital (Other); The Second People's Hospital of Huai'an (Other); The Third People's Hospital of Kunshan (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAC-HAAG-02
Record Dates: First submitted 2019-09-08; First posted 2019-09-10 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Acute Myeloid Leukemia; Induction Chemotherapy
Keywords: Decitabine, HAAG, AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Decitabine; Homoharringtonine; Aclarubicin; Cytarabine; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Decitabine combined with HAAG Regimen (Experimental): This cohort will determine the safety and efficacy of decitabine combined with HAAG regimen in elderly newly diagnosed AML patients.
  Interventions: Drug: Decitabine, Homoharringtonine, Aclarubicin, Cytarabine and G-CSF

INTERVENTIONS:
Drug: Decitabine, Homoharringtonine, Aclarubicin, Cytarabine and G-CSF — Decitabine:20mg/m2/d, d1~5, intravenous infusion; Homoharringtonine:1mg/d,d3~9,intravenous infusion; Aclarubicin:10mg/d, d3~d6, intravenous infusion; Cytarabine:10mg/m2,q12h,d3-9, subcutaneous injection;
  Granulocyte colony-stimulating factor:
  50-300μg/d (when WBC counts are less than 20×10^9/L ),subcutaneous injection;

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of DAC combined with HAAG regimen in the induction treatment of newly diagnosed AML patients older than 60 years.

DETAILED DESCRIPTION:
This is a phase 3, open Label, single arm, multi-center study in elderly newly diagnosed AML patients. The patients will receive DAC combined with HAAG in the induction treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed AML according to the WHO (2016) classification of acute myeloid leukemia.
2. 60-79 years old.
3. ECOG score: 0-3.
4. No history of previous chemotherapy or target therapy.
5. Provide informed consent.

Exclusion Criteria:

1. Patients have acute promylocytic leukemia or chronic myeloid leukemia in blast crisis.
2. Patients with another malignant disease.
3. Patients with uncontrolled active infection.
4. Patients with left ventricular ejection fraction < 0.5 by echocardiography or grade III/IV cardiovascular dysfunction according to the New York Heart Association Classification.
5. Patients with aspartate aminotransferase or glutamic-pyruvic transaminase > 3x upper limit of normal or bilirubin > 2.0 mg/dL.
6. Patients with creatinine clearance rate < 50ml/min.
7. Patients with active hepatitis B or hepatitis C infection.
8. Patients with HIV infection.
9. Patients with other commodities that the investigators considered not suitable for the enrollment.

Ages: 60 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Day 28-35 of induction course
  ORR includes complete response (CR), CRi and PR. CR was defined as < 5% bone marrow blasts in an aspirate with spicules, no blasts with Auer rods or persistence of extramedullary disease, and independent of transfusions; CRi: was defined as<5% bone marrow blasts, either ANC<1×10^9/L or platelets<100×10^9/L, transfusion independence but with persistence of cytopenia; PR was defined as decrease of at least 50% in the percentage of blasts to 5-25% in the bone marrow aspirate and the normalization of blood counts.

SECONDARY OUTCOMES:
Overall survival (OS) | 3 years
  time from randomization to death from any cause
Leukemia-free survival (LFS) | 3 years
  time from randomization to the first relapse or death
Cumulative incidence of relapse (CIR) | 3 years
  time from achievement of a remission to the first relapse
Number of adverse events | 2 years
  adverse events are evaluated with CTCAE V5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaowen Tang, Ph.D., Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- the First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China